CLINICAL TRIAL: NCT03221985
Title: Investigating the Relationship Between Mobile Phone Usage and Emotions. A Pilot Study Using the Experienced Sampling Method
Brief Title: ESM Pilot: Mobile Phones and Psychology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL55632.068.15
Record Dates: First submitted 2017-05-14; First posted 2017-07-19 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Communication; Addiction; Affect
Keywords: experience sampling method
MeSH Terms: conditions — Communication; Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Questionnaires (Other)
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — questionnaire with application on smartphone

SUMMARY:
The research team will investigate whether there is a relation between smartphone usage and psychological parameters using the smartphone application.

DETAILED DESCRIPTION:
There are indications for mobile phone effects on psychological and psychological functioning. Most publications on this subject report effects on 'mobile phone addiction'. A methodological problem in these studies is the collection of data in retrospect. With the mobile phone application it is possible to prevent this type of bias. By collecting real-life data in a longitudinal design with a 2 x N=1 pilot study, it is possible to obtain an impression of the relationship between mobile phone usage and emotion/behavior efficiently.

The objective of this study is to investigate whether there is a relation between smartphone usage and psychological parameters in young adults. Taking into accordance the type of research (observational) and the present state of literature (the relationship between mobile phones and psychological effects has not been studied before using the experience sampling method (E.S.M.)) the following hypothesis are formulated. It is expected that the undesired absence of one's phone will lead to an enlarged stress level. Furthermore, it is expected that an increase of phone usage will lead to more depressive symptoms, to less concentration and to sleep disturbance. Finally, it is expected that loneliness will lead to increased phone usage.

A longitudinal pilot study, in which the participant will be asked to fill out the mobile phone application questionnaire 10 times a day at random moments on a smartphone, during a 3 months period.

The mobile phone application questionnaire contains a series of multiple choice questions about the present affect (three positive, five negative), the present context and activities (physical activity, occupation, presence of other people), physical discomfort (fatigue, concentration level, pain) and mobile phone usage (frequency, frustration when unable to use phone) since the last beep. Positive affect: cheerful, mentally fit and relaxed. Negative affect: irritated, bored, lonely, stressed and worrying. The answers will be registered using a 7-point Likert scale, ranging from 'not' to 'very'.

Participants will be invited to the research location twice for a briefing (30 minutes) and a debriefing session (30 minutes). Furthermore the participants will be asked to fill out the mobile phone application questionnaire on a daily base after every beep. It is expected this will cost a time investment of approximately 15 minutes per day. The questionnaires are generally experienced as a small burden (in previous research performed by this department). Participation is not associated with health risks.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* good understanding of dutch language
* smartphone user

Exclusion Criteria:

* psychiatric diagnosis
* pregnancy

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire using the experience sampling method, administered by the mobile phone application. | after 3 months
  The mobile phone application questionnaire will be offered 10 times a day at random moments on the smartphone of the participants, during a 3 months period.
  The mobile phone application questionnaire contains a series of multiple choice questions about the present affect (three positive, five negative), the present context and activities (physical activity, occupation, presence of other people), physical discomfort (fatigue, concentration level, pain) and mobile phone usage (frequency, frustration when unable to use phone) since the last beep. Positive affect: cheerful, mentally fit and relaxed. Negative affect: irritated, bored, lonely, stressed and worrying. The answers will be registered using a 7-point scale, ranging from 'not' to 'very'.

CONTACTS AND LOCATIONS:
Overall Officials: Jim van Os, prof. dr., Principal Investigator — Maastricht University
Locations (1):
- Mondriaan, locatie Vijverdal, Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
digitally obtained data will be uploaded

REFERENCES:
- [Derived] Roggeveen S, van Os J, Bemelmans K, van Poll M, Lousberg R. Investigating Associations Between Changes in Mobile Phone Use and Emotions Using the Experience Sampling Method: Pilot Study. JMIR Form Res. 2018 Jun 18;2(1):e12. doi: 10.2196/formative.8499. PMID 30684428